CLINICAL TRIAL: NCT04636775
Title: Microbiome in Immunotherapy naïve NSCLC Patients Receiving PD-1/L1 Blockade (MIP_NSCLC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jun Zhang, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, MD, PhD, Associate Professor; Principal Investigator, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: IIT-2020-MIP-NSCLC
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: NSCLC Stage IV; NSCLC, Recurrent
Keywords: Advanced NSCLC; Metastatic NSCLC; Recurrent NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Microbiota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal and buccal swabs, and stool sample, as well as the extracted DNAs for current and future, study-related research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunotherapy naïve NSCLC patients: Microbiome in immunotherapy naïve NSCLC patients receiving PD-1/L1 blockade
  Interventions: Diagnostic Test: Microbiome

INTERVENTIONS:
Diagnostic Test: Microbiome — Nasal and buccal swabs, and stool sample, as well as the extracted DNAs

SUMMARY:
This phase IV study is hoping to determine if examining the microbiome in non-small cell lung cancer, immunotherapy naive participants can predict the effectiveness of immunotherapy treatment as well as determine ahead of time adverse events and their severity. In addition, the investigator will look into microbiome changing modifiers.

ELIGIBILITY:
Inclusion Criteria:

* Must have tumor tissue biopsy-proven to be NSCLC
* Must have a target lesion to evaluate treatment response
* Immunotherapy naïve metastatic/advanced/recurrent NSCLC patients
* Will receive single agent anti-PD-1/PD-L1 therapy (e.g. pembrolizumab, nivolumab, atezolizumab, avelumab or durvalumab, etc.). Patients can be on other interventional trial if they will be receiving single agent anti-PD-1/PD-L1

Exclusion Criteria:

* Prior treatment with any forms of cancer immunotherapy
* Not competent to make medical decision, noncommunicative or noncompliant per treating physician's judgement
* Not English-speaking
* Patients that are pregnant
* Prisoners
* Students and employees
* Psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Immunotherapy naïve metastatic/advanced/recurrent NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome difference between patients with and without AEs>=grade 3 | Through study completion, an average of 1 year
  Adverse events (AEs) will be graded per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Microbiome difference between responders vs. nonresponders | Through study completion, an average of 1 year
  Treatment response will be evaluated using the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1
Correlation of microbiome to tumor tissue PD-L1 expression | Through study completion, an average of 1 year
  PD-L1 expression is per standard of care using IHC
Correlation of microbiome to diet | Through study completion, an average of 1 year
  Customized Diet Survey

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Principal Investigator — The University of Kansas Cancer Center
Locations (3):
- United States (3):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swami U, Zakharia Y, Zhang J. Understanding Microbiome Effect on Immune Checkpoint Inhibition in Lung Cancer: Placing the Puzzle Pieces Together. J Immunother. 2018 Oct;41(8):359-360. doi: 10.1097/CJI.0000000000000232. PMID 29781826
- [Background] Strouse C, Mangalam A, Zhang J. Bugs in the system: bringing the human microbiome to bear in cancer immunotherapy. Gut Microbes. 2019;10(2):109-112. doi: 10.1080/19490976.2018.1511665. Epub 2018 Sep 5. PMID 30183502